CLINICAL TRIAL: NCT06685159
Title: Risk Factors for Postoperative Complications in Surgery With Pneumoperitoneum in Trendelenburg Position. Observational Pilot Study
Brief Title: Predictors of Postoperative Complications in Surgery With Pneumoperitoneum in the Trendelenburg Position
Status: Recruiting | Type: Observational
Sponsor: Reuven Pizov (Other)
Responsible Party: Sponsor-Investigator, Reuven Pizov, Anesthesia Department Chair, Hadassah Medical Organization
Organization: Hadassah Medical Organization (Other)
Other Study IDs: 0303-23 HMO
Record Dates: First submitted 2024-11-06; First posted 2024-11-12 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Trendelenburg Position; Pneumoperitoneum
MeSH Terms: conditions — Pneumoperitoneum | interventions — Laparoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and urine samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Procedure: Laparoscopic Surgery — Laparoscopic surgery (with controlled pneumoperitoneum) in the Trendelenburg position

SUMMARY:
Evaluate early postoperative complications after surgery in Trendelenburg position with increased intraabdominal pressure (surgery with pneumoperitoneum). Evaluate the relationship between hemodynamic and metabolic changes on perioperative outcome.

ELIGIBILITY:
Inclusion Criteria:

* ASA Class I-IV.
* Planned for laparoscopic surgery in the Trendelenburg position that is expected to last more than 2 hours.
* Planned arterial catheter insertion.

Exclusion Criteria:

* Pregnancy.
* Planned open abdominal surgery.
* Renal Replacement Therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients who undergo elective laparoscopic surgery in the Hadassah Ein-Kerem Medical Center
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-06-19 (Actual); Primary Completion 2026-06-19 (Estimated); Study Completion 2026-06-19 (Estimated)

PRIMARY OUTCOMES:
Perioperative change in urine NGAL | Baseline (after anesthesia induction but before beginning of surgery) and 2h hours after completion of surgery
  Measurement of the concentration of neutrophil gelatinase-associated lipocalin (as an early marker of kidney injury) in a urine sample taken from a Foley catheter
Acute Kidney Injury | 2 hours after completion of surgery; 1 day after the procedure; 3 days after the procedure.
  According to the KDIGO acute renal injury stage
Perioperative change in serum NGAL | Baseline (after anesthesia induction but before beginning of surgery) and 2h hours after completion of surgery
  Measurement of the concentration of neutrophil gelatinase-associated lipocalin (as an early marker of kidney injury) in a blood sample
Perioperatitve change in serum concentration of Cannabidiol | Baseline (after anesthesia induction but before beginning of surgery) and 2h hours after completion of surgery and 2h hours after completion of surgery
  Measurement of the concentration of cannabidiol (as an early marker of kidney injury) in a blood sample
Perioperatitve change in urine concentration of Cannabidiol | Baseline (after anesthesia induction but before beginning of surgery) and 2h hours after completion of surgery
  Measurement of the concentration of cannabidiol (as an early marker of kidney injury) in a urine sample taken from a Foley catheter
Perioperatitve change in TBW | Baseline (after anesthesia induction but before beginning of surgery) and 2h hours after completion of surgery
  Perioperative change in the bioimpedence-based measurement of Total Body Water (TBW)
Perioperatitve change in ECW | Baseline (after anesthesia induction but before beginning of surgery) and 2h hours after completion of surgery
  Perioperative change in the bioimpedence-based measurement of Extracellular Water (ECW)
Perioperatitve change in serum pH | Baseline (after anesthesia induction but before beginning of surgery) and 2h hours after completion of surgery
  As measured by arterial blood gas
Perioperatitve change in serum BE | Baseline (after anesthesia induction but before beginning of surgery) and 2h hours after completion of surgery
  Perioperatitve change in serum Base Excess (BE) As measured by arterial blood gas
Perioperatitve change in serum lactate concentration | Baseline (after anesthesia induction but before beginning of surgery) and 2h hours after completion of surgery
  Perioperatitve change in serum lactate concentration as measured by arterial blood gas
Perioperatitve change in serum syndecan-1 concentration | Baseline (after anesthesia induction but before beginning of surgery) and 2h hours after completion of surgery
  Measured by ELISA

SECONDARY OUTCOMES:
Delirium | Within 7 days after surgery
  As assessed by CAM-ICU
CVA / TIA | Within 30 days after surgery
  New diagnosis of cerebrovascular accident or transient ischemic attack
Myocardial Ischemia | During hospital stay, within 30 days after surgery
  New myocardial ischemia, as diagnosed by ecg or serum troponin
Arrhythmia | During hospital stay, within 30 days after surgery
  New clinically significant arrhythmia
Atelectasis | During hospital stay, within 30 days after surgery
  New atelectasis
Pneumonia | During hospital stay, within 30 days after surgery
  According to CDC criteria
ARDS | During hospital stay, within 30 days after surgery
  New Acute Respiratory Distress Syndrome (ARDS) according to Berlin criteria

CONTACTS AND LOCATIONS:
Locations (1):
- Hadassah Medical Center, Jerusalem, Yerushalaim, Israel